CLINICAL TRIAL: NCT03179878
Title: A Phase 1, First-in-human, Oral Single and Multiple Dose-Escalation, Randomized, Double-blinded, Placebo-controlled Study of SYNB1020 in Healthy Adult Volunteers to Evaluate Safety, Tolerability, Dosing, and Pharmacodynamics
Brief Title: Safety and Tolerability of SYNB1020-CP-001
Acronym: SYNB1020CP001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYNB1020-CP-001
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteer; Urea Cycle Disorder
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blinded, Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SYNB1020 (Experimental): SYNB1020
  Interventions: Drug: SYNB1020
- Placebo (Placebo Comparator): 100 mL masking solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: SYNB1020 — Investigational Product
  Arms: SYNB1020

SUMMARY:
A Phase 1, First-in-human, Oral Single and Multiple Dose-Escalation, Randomized, Double-blinded, Placebo-controlled Study of SYNB1020 in Healthy Adult Volunteers to Evaluate Safety, Tolerability, Dosing, and Pharmacodynamics

DETAILED DESCRIPTION:
This Phase 1, dose-escalating, randomized, double-blinded study will evaluate SYNB1020 in placebo-controlled cohorts within the following 2 study parts:

Part 1: A single-ascending dose (SAD) study conducted in an inpatient setting over 6 days in healthy volunteer male and female subjects evaluated in up to 7 dose cohorts to identify the maximum tolerated dose (MTD) within the single dose range studied; and Part 2: A multiple-ascending dose (MAD) study conducted in an inpatient setting over 22 days in healthy volunteer male and female subjects evaluated in up to 4 dose cohorts that were proven tolerable in the SAD part of the study to identify the MTD of SYNB1020 within the multiple-dose range studied. Up to 48 subjects may be enrolled in this part of the study.

Subjects will be screened for eligibility within 30 days prior to enrollment, with evaluations of exercise habits, gastrointestinal (GI) signs and symptoms, fecal patterns (frequency, consistency), recent or current antibiotic exposure, and laboratory measurements. Eligible patients will be admitted to an inpatient facility for investigational product (IP) administration, safety monitoring, and collection of blood, urine, and fecal samples for pharmacokinetic and pharmacodynamic evaluations.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 to 64 years
* Healthy volunteer Males and Females; Females must be of non childbearing potential
* Able and willing to complete informed consent process
* Available for and agree to all study procedures
* Screening Labs within normal range

Key Exclusion Criteria:

* Acute or chronic medical, surgical, psychiatric, social or laboratory abnormality
* Body mass index < 18.5 or ≥ 30 kg/m2
* Intolerance of or allergic reaction to E. coli Nissle or any of the ingredients in SYNB1020 or placebo formulations; allergies to common foods (e.g., eggs, milk, soy, nuts).
* Prior participation in a study with SYNB1020
* Evidence or history of clinical signification hematological, renal, endocrine, pulmonary, GI cardiovascular, hepatic, psychiatric, neurologic or allergic disease
* Personal or family history of UCD

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events, Laboratory Assessments and ECGs to measure Safety and Tolerability of SYNB1020 | 3 months from study entry
  Will be measured by assessing nature and frequency of AEs, Laboratory Assessments, and ECGs

SECONDARY OUTCOMES:
GI tolerability measured using the Gastrointestinal Symptom Rating Scale (GSRS) | 1 month of study entry
  Will be measured using the Gastrointestinal Symptom Rating Scale (GSRS)
SYNB1020 kinetics measured by qPCR fecal assays | 3 months from study entry
  Will be measured by qPCR fecal assays

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: No